CLINICAL TRIAL: NCT06240520
Title: Optimizing Reversal of HIV Latency With Combination Therapy (Pyrimethamine, Lenalidomide, Panobinostat)
Brief Title: Optimizing Reversal of HIV Latency With Combination Therapy
Acronym: ORBIT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); AIDSfonds (Unknown)
Responsible Party: Principal Investigator, Casper Rokx, associate professor, internist and infectious diseases specialist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-511192-15-00
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Hiv
Keywords: HIV Cure; Shock and kill; Latency reversal; Combination therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Shock | interventions — Panobinostat; Pyrimethamine; Tablets; Lenalidomide

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- control (No Intervention)
- panobinostat (Experimental)
  Interventions: Drug: Panobinostat 20 MG Oral Capsule
- lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide 25 MG Oral Capsule
- pyrimethamine (Experimental)
  Interventions: Drug: Pyrimethamine 200mg Oral Tablet
- panobinostat + lenalidomide (Experimental)
  Interventions: Drug: Panobinostat 20 MG Oral Capsule; Drug: Lenalidomide 25 MG Oral Capsule
- panobinostat + pyrimethamine (Experimental)
  Interventions: Drug: Panobinostat 20 MG Oral Capsule; Drug: Pyrimethamine 200mg Oral Tablet
- lenalidomide + pyrimethamine (Experimental)
  Interventions: Drug: Pyrimethamine 200mg Oral Tablet; Drug: Lenalidomide 25 MG Oral Capsule

INTERVENTIONS:
Drug: Panobinostat 20 MG Oral Capsule — Panobinostat 20mg will be administered once orally
  Arms: panobinostat; panobinostat + lenalidomide; panobinostat + pyrimethamine
Drug: Pyrimethamine 200mg Oral Tablet — Pyrimethamine 200mg will be administered once orally
  Arms: lenalidomide + pyrimethamine; panobinostat + pyrimethamine; pyrimethamine
Drug: Lenalidomide 25 MG Oral Capsule — Lenalidomide 25mg will be administered once orally
  Arms: lenalidomide; lenalidomide + pyrimethamine; panobinostat + lenalidomide

SUMMARY:
The ORBIT trial is part of a worldwide search for a functional cure of HIV. One such cure strategy aims to reverse HIV in the reservoir from latency by increasing cell-associated HIV-RNA, which will lead to increased antigen presentation, trigger immune recognition, and facilitate the elimination of reservoir cells (so-called 'shock and kill' approach to HIV cure). Participants of the trial are adults with HIV with undetectable viral load that are able to give informed consent to participate in the trial, in total 49 patients will be recruited. The investigational medical compounds in this trial are panobinostat, lenalidomide and pyrimethamine. These are all licensed drugs for other conditions. Participants of this trial will receive a single dose of the IMPs, either as monotherapy or as combination therapy. Sampling will be performed before, during and after medical treatment to evaluate latency reversal, reservoir reduction and safety endpoints. Patients will be recruited from the Erasmus MC, Amsterdam university Medical Center and the University Medical Center Utrecht.

DETAILED DESCRIPTION:
Rationale

Despite advances in antiretroviral therapy (ART) that nowadays can fully suppress HIV replication, HIV treatment still has to be taken lifelong due to the persistence of a latent HIV reservoir. This reservoir consists of long-lived memory T-cells in which HIV persists as provirus in the host genome. There is minimal proviral transcriptional activity, and the elimination of these reservoir cells is prohibited by limited antigen recognition and elimination by the immune system. When antiretroviral treatment is stopped, the virus almost universally rebounds from its reservoir, and if left untreated will result in HIV disease progression. Intensive research efforts over the last decade is focused on finding a definitive cure for HIV that would allow people to safely stop their ART without risking viral rebound. One such cure strategy aims to reverse HIV in the reservoir from latency by increasing cell-associated HIV-RNA, which will lead to increased antigen presentation, trigger immune recognition, and facilitate the elimination of reservoir cells (so-called 'shock and kill' approach to HIV cure). Several latency reversal agents have been identified to reactivate HIV transcription in the reservoir. Though current single latency reversal agents are effective in achieving this to a limited extent, they have not resulted in significant HIV reservoir reduction. One explanation could be that a stronger reactivation is needed. As such, we aim to study novel combinations of promising latency-reversing agents with different drug targets to improve HIV latency reversal within the viral reservoir.

Study design:

Open label randomized controlled trial.

Study population:

49 adult people with HIV-1

Intervention:

The investigational drugs are panobinostat, lenalidomide, and pyrimethamine. Patients will be randomized 1:1:1:1:1:1:1 to one of 7 arms to receive a combination of two investigational drugs, one investigational drug or no interventional treatment.

Arm 1: control Arm 2: panobinostat 20mg once orally Arm 3: lenalidomide 25mg once orally Arm 4: pyrimethamine 200mg once orally Arm 5: panobinostat 20mg once orally and lenalidomide 25mg once orally. Arm 6: panobinostat 20mg once orally and pyrimethamine 200mg once orally. Arm 7: lenalidomide 25mg once orally and pyrimethamine 200mg once orally.

Procedures

All participants will have a screening visit including a leukapheresis or venous blood sampling before the intervention between T= -1 to -60 days. Subsequent blood sampling by phlebotomy is at T=0-hour (day 0) before drug administration, and T=2 hours, T=6 hours, T=24 hours (day 1), and T= 2 months (60 days) post study drug administration. An optional second leukapheresis instead of blood sampling by phlebotomy at the last sampling time point is possible. Clinical assessments are at days 0, 1, and 7. Clinical assessment at day 7 can optionally be remote.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection by 4th generation ELISA, Western Blot or PCR.
* ≥ 18 years old.
* World Health Organization (WHO) performance status 0 or 1.
* Current plasma HIV RNA <50 copies/ml measured on the last 2 occasions, with measurements being at least 3 months apart.
* Uninterrupted prescribed ART for a minimum of two consecutive years.
* Considered >95% adherent to ART by treating physician.
* Current blood CD4+T-cell count of ≥200 cells/mm3
* No clinical signs of cellular immunodeficiency or AIDS.
* Pre-ART plasma HIV RNA ≥1000 copies/mL.
* Confirmed HIV subtype B. People with a high likelihood of subtype B can participate if they live in a HIV subtype B endemic region with HIV acquired there and in whom no HIV sequencing is available or can be done on stored samples.
* People should be considered capable mentally and somatically by their treating physician to understand the informed consent procedure and undergo the study treatment.

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:
* Previous exposure to any of the studied LRAs in the last year
* Acute or chronic co-infection with hepatitis B and/or C by the presence of hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA in blood.
* Co-medication with clinically significant interactions with LRA (see chapter 15.h for list)
* Comorbidities affected by LRA compounds, such as but not limited to: known Glucose-6-phospate-dehydrogenase (G6PD) deficiency with anaemia, untreated haemolysis of any cause or hereditary thrombophilia not currently treated by anticoagulation.
* Prolonged Qtc time >480ms at screening, as measured by electrocardiogram (ECG).
* Patients of childbearing potential unless double contraceptive measures are taken. Non-childbearing is defined by one of the following criteria: amenorrhoea for ≥ 1 year, premature ovarian failure, assigned male at birth, or having undergone previous bilateral salpingo-oophorectomy, or hysterectomy
* Sexual active patients unwilling to abstain from sex unless willing to use condom protection during and until 1 week after administration of study medication.
* Active malignancy during the past year with the exception of basal carcinoma of the skin, stage 0 cervical carcinoma, Kaposi's sarcoma treated with ARTalone or other indolent malignancies.
* Registered allergies for any of the investigational medical products
* Any lab abnormalities at screening as listed below:
* Moderate kidney impairment, defined as eGFR <50 mL/min
* Moderate hepatic impairment, defined as bilirubin > 3 x upper limit of normal (ULN) or ALT > 3x ULN
* Inadequate blood counts, defined as: Haemoglobin <6.5 mmol/L (males) or <6.0 mmol/L (females), absolute neutrophil count <1000 cells/mm3, thrombocytes <100 x109/L, international standardized ratio >1.6, activated partial thromboplastin time >40 seconds, serum sodium <130 mmol/L, serum potassium <3.0 mmol/L, serum phosphate <0.5 mmol/L, serum calcium <1.9 mmol/L, serum magnesium <0.5 mmol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Cell-associated HIV RNA | 1 day
  Fold change in cell-associated HIV RNA
Adverse events | 14 days
  The number and severity of clinical and biochemical adverse events considered by the investigator to be related to any of the investigational drugs

SECONDARY OUTCOMES:
HIV reservoir | 120 days
  The change in the HIV reservoir size and genetic composition from baseline to the end of the study

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Erasmus Medical Centre, Rotterdam, South Holland
  - Amsterdam University Medical Center, Amsterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored under FAIR use principle for use in future research. Should external researchers want to use this dataset, they can contact the principal investigator. In the case of adequate privacy standards data can be shared under a specific new Data Sharing Agreement
Supporting Information: SAP, Analytic Code
Time Frame: Data will be available after publication of primary results. Data will kept in storage for 15 years
Access Criteria: Receiving facility has data privacy protection meeting EU GDPR standards